CLINICAL TRIAL: NCT05385978
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Parallel-group Proof-of-concept Study to Evaluate Efficacy and Safety of Distal Jejunal-release Dextrose (Aphaia Technology, AT) in Obese Subjects
Brief Title: A Study of Distal Jejunal-release Dextrose in Obese Participants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aphaia Pharma US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 034B20
Record Dates: First submitted 2022-05-13; First posted 2022-05-23 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Obese
Keywords: Obese; Dextrose; Hypertension; NASH; 034B20; Distal jejunal-release dextrose; Endocrine disorders; Metabolic conditions; NAFLD
MeSH Terms: conditions — Obesity; Hypertension; Endocrine System Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized, double-blind, placebo-controlled, parallel-group proof-of-concept efficacy and safety study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APHD-012 (Active Comparator): Participants will receive a single dose of APHD-012 12 g daily, under fasting conditions prior to main daily meals for 180 days (6 months) for Cohort 2 and for 360 days (12 months) for Cohort 1.
  Interventions: Drug: APHD-012
- APHD-012P (Placebo Comparator): Participants will receive a single dose of APHD-012P daily, under fasting conditions prior to main daily meals for 180 days (6 months) for Cohort 2 and for 360 days (12 months) for Cohort 1.
  Interventions: Drug: APHD-012P

INTERVENTIONS:
Drug: APHD-012 — Distal jejunal-release dextrose beads (Aphaia technology, AT)
  Other Names: Distal jejunal-release dextrose beads
  Arms: APHD-012
Drug: APHD-012P — Distal jejunal-release placebo beads
  Other Names: Placebo
  Arms: APHD-012P

SUMMARY:
The primary purpose of the study is to evaluate the efficacy and safety of APHD-012 (distal jejunal-release dextrose [Aphaia technology, AT]) in obese participants.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, phase II proof-of-concept study to be conducted in 150 adult obese male and female participants who are 18 to 70 years of age with or without one or more endocrine and/or metabolic conditions. The study aims to evaluate the efficacy and safety of distal jejunal-release dextrose (Aphaia technology, AT) in obese participants.

Participants will be randomly assigned to receive either APHD-012 (distal jejunal-release dextrose or APH-012P (a matching placebo). There will be two cohorts in the study. Participants from Cohort 1 will receive study medication once daily for 12 months (360 days), and participants from Cohort 2 will receive study medication once daily for 6 months (180 days).

Overall, 150 participants will be enrolled in the study:

* Cohort 1 (60 participants) - 6-month treatment period + 6-month maintenance treatment period
* Cohort 2 (90 participants) - 6-month treatment period

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 30.0-39.9 kg/m^2 and/or waist circumference: men >102 cm, women >88 cm
* Stable body weight: gain or loss in body weight ≤5 kg over last 3 months
* Obese participants with or without one or more of the following conditions:

  1. NAFLD - simple steatosis based on a FibroScan CAP™ test result at screening (CAP Score ≥238 decibel-milliwatts (dB/m) (Steatosis Grades 1-3) with no or mild fibrosis (F0-F1 fibrosis Score)
  2. NASH - steatohepatitis based on FibroScan fibrosis Score at screening (≥7.5 kPa and <14 kPa (Stage F2-F3)
  3. Confirmed medical history of metabolic syndrome
  4. Homeostatic Model Assessment of Insulin Resistance (HOMA IR) Score ≥2
  5. Confirmed medical history of type 2 diabetes mellitus (T2DM) diagnosis or HbA1c ≥7.0 and <11 (based on screening values)
  6. High total cholesterol ≥240 mg/dL (based on screening values)
  7. Hypertension (participants with Stage 1 hypertension (systolic blood pressure [SBP] ≥130 mmHg <180 mmHg, diastolic blood pressure [DBP] ≥80 mmHg <110 mmHg) (based on screening values)
* If on medication to manage endocrine/metabolic conditions, must be on stable doses of medication ≥3 months prior to screening:

  1. Participants with T2DM may be treated with either diet and exercise alone, metformin, sulphonylurea, thiazolidinediones, sodium-glucose cotransporter-2 (SGLT-2) inhibitors, and bromocriptine quick-release (QR) as single agents or combination therapy.
  2. As lipid-lowering medication participants may be treated with statins and fibrates, proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors, ezetimibe, or supplements like omega-3-fatty acids.
  3. As antihypertensive medication participants may be treated with beta-blockers, angiotensin-converting enzyme (ACE) inhibitors, angiotensin-II-inhibitors, diuretics, or calcium channel blockers.
* Normal GI function, or abnormalities which the clinical investigator does not consider a disqualification for participation in the study

Exclusion Criteria:

* Incomplete Coronavirus Disease of 2019 (COVID-19) vaccination
* Treatment with weight loss medications in the past 3 months
* Proven history of bulimia or anorexia nervosa
* Treatment with injectable antidiabetic medications in the last 3 months (e.g. Glucagon-like peptide-1 [GLP-1] receptor agonists, insulin)
* Treatment with dipeptidyl peptidase-4 inhibitors in the last 3 months
* NASH with cirrhosis (fibrosis Score=F4 (≥14 kPa) as determined by screening FibroScan
* Confirmed medical history of liver cirrhosis, cholestatic disease, alcohol-related liver disease
* Type 1 diabetes mellitus, HbA1c ≥11, fasting plasma glucose levels ≥270 mg/dL
* Proliferative retinopathy or maculopathy
* Abnormal liver function tests:

  1. Transaminases:

     * Alanine transaminase (ALT)/aspartate aminotransferase (AST) ≥5 x upper limit of normal (ULN) for participants with NAFLD or NASH (as determined by screening FibroScan)
     * ALT/AST ≥2.5 x ULN for participants without NAFLD or NASH (as determined by screening FibroScan)
  2. Alkaline phosphatase (ALK) ≥2.5 x ULN
  3. Total bilirubin ≥2 x ULN
* Stage 4 hypertension (SBP ≥180, DBP ≥110)
* History or presence of any uncontrolled cardiovascular, pulmonary, hepatobiliary, renal, hematologic, gastrointestinal, endocrinologic, immunologic, dermatologic, neurological, psychiatric, metabolic, musculoskeletal, or malignant disease (except conditions accepted for inclusion) which the clinical investigator does not consider a disqualification for participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-11 (Estimated); Study Completion 2024-11-11 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline in Percent Weight Change Compared with Placebo | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Bodyweight measurements will be done using standard personal balance referring to kilogram-Scale. Weighing will be done without shoes and with just underwear on. It is important that weighing is always done in the same way, preferably in the morning, before eating or drinking.

SECONDARY OUTCOMES:
Percentage of Participants with ≥2.5% Baseline Body Weight Loss at 6 Months Compared with Placebo (Weight Loss Responders) | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Body weight measurements will be done using standard personal balance referring to kilogram-Scale. Weighing will be done without shoes and with just underwear on. It is important that weighing is always done in the same way, preferably in the morning, before eating or drinking.
Percentage of Participants with ≥5% Baseline Body Weight Loss at 6 Months Compared with Placebo (Weight Loss Responders) | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Body weight measurements will be done using standard personal balance referring to kilogram-Scale. Weighing will be done without shoes and with just underwear on. It is important that weighing is always done in the same way, preferably in the morning, before eating or drinking.
The Difference in Mean Absolute Weight Loss Compared with Placebo at 6 Months | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Body weight measurements will be done using standard personal balance referring to kilogram-Scale. Weighing will be done without shoes and with just underwear on. It is important that weighing is always done in the same way, preferably in the morning, before eating or drinking.
Mean Absolute Change and Percent Change of Waist Circumference | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Waist circumference measurements will be done using a standard measuring tape referring to centimeter Scale.
Mean Absolute Change and Percent Change of Systolic Blood Pressure and Diastolic Blood Pressure | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be measured using a standard sphygmomanometer with the Riva-Rocci cuff and a stethoscope; alternatively, an automatic device with upper arm cuff can be used. Measurements are done in sitting position after 5 minutes of rest.
Mean Absolute Change and Percent Change of Heart Rate | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Heart rate measurement will be obtained along with the blood pressure measurement.
Mean Absolute Change and Percent Change of Triglycerides and Cholesterol | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Triglycerides and cholesterol (including total cholesterol, low-density lipoprotein [LDL], and high-density lipoprotein [HDL]) will be measured using standard clinical laboratory methods at the site laboratories.
Mean Absolute Change and Percent Change of Homeostatic Model Assessment of Insulin Resistance | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Homeostasis model assessment-estimated insulin resistance (HOMA-IR) will be determined with standard clinical laboratory methods.
Mean Absolute Change and Percent Change of Fasting Plasma Glucose, Fasting Plasma Insulin and Glycated Hemoglobin | At Baseline and at each visit until Day 180 for Cohort 2 and Day 360 for Cohort 1
  Fasting plasma glucose will be determined using a standard blood glucometer. Fasting plasma insulin will be determined with standard clinical laboratory methods. Glycated hemoglobin (HbA1c) will be measured using a standard enzyme-linked immunoassay (ELISA) method.
  HbA1c will be measured in participants with type two diabetes (T2DM).
Mean Absolute Change and Percent Change of Alanine Transaminase, Aspartate Transaminase and Gamma Glutamyl Transpeptidase | At Baseline and at Day 90, at Day 180 for Cohort 2 and at Day 360 for Cohort 1
  Liver enzymes (ALT, AST, GGT) will be measured using standard clinical laboratory methods.
Mean Absolute Change and Percent Change of Fatty Liver Controlled Attenuation Parameter Score and Liver Fibrosis Score | At Baseline and at Day 90, at Day 180 for Cohort 2 and at Day 360 for Cohort 1
  Fatty liver Controlled Attenuation Parameter (CAP) Score will be measured in:
  * Participants with Non-alcoholic fatty liver disease (NAFLD): Steatosis grade and;
  * Participants with Non-alcoholic steatohepatitis (NASH): fibrosis Score category
  Fatty liver CAP Score and liver fibrosis Score will be measured using FibroScan™ equipment or equivalent.
Number of Participants Reported with At least One Treatment Emergent Adverse Event (TEAE) | At each visit until Day 180 for Cohort 2 and until Day 360 for Cohort 1
  A treatment-emergent adverse event is defined as any event not present prior to the initiation of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment
Advance Understanding of Dose/Exposure - Response Relationships | At Baseline, at Day 90, Day 180 and at Day 360 for Cohort 1
  Dose/Exposure - Response Relationships will be evaluated.

OTHER OUTCOMES:
Glucagon-like Peptide-1 Level Determination | At Baseline, at Day 90, Day 180 and at Day 360 for Cohort 1
  Blood samples of 2 mL will be taken at pre-dose (-0.5 h [within 5 minutes]) and 1.0, 2.0, 3.0, 4.0, 5.0, 6.0 and 8.0 hours after investigational medicinal product administration.
  The blood samples for the determination of Glucagon-like peptide-1 (GLP-1) and circulating biomarkers and micro Ribonucleic acid (miRNA)1983 will be collected in BD P800 tubes.
Area Under the Plasma Concentration-time Curve from Time 0 to 8 Hours (AUC0-8) | At Baseline, at Day 90, Day 180 and at Day 360 for Cohort 1
Maximum Plasma Concentration (Cmax) | At Baseline, at Day 90, Day 180 and at Day 360 for Cohort 1
Time to Reach the Maximum Plasma Concentration (Tmax) | At Baseline, at Day 90, Day 180 and at Day 360 for Cohort 1

CONTACTS AND LOCATIONS:
Locations (9):
- Georgia (5):
  - LTD "Israeli-Georgian Medical Research Clinic Healthycore", Tbilisi
  - LTD "Acad. G. Chapidze Emergency Cardiology Center", Tbilisi
  - LTD "Diacor", Tbilisi
  - LTD "National Institute of Endocrinology", Tbilisi
  - LTD "Tbilisi Heart Center", Tbilisi
- Germany (2):
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Ruppin-Brandenburg, Neuruppin
- Puerto Rico (2):
  - GCM Medilcal Group, San Juan
  - FDI Clinical Research, San Juan

IPD SHARING:
Plan to Share IPD: No